CLINICAL TRIAL: NCT06285877
Title: Study on the Effectiveness of the Use of the Nintendo Switch Combined With Conventional Therapy in People With Acquired Brain Injury: A Pilot Study
Brief Title: Effectiveness of the Use of the Nintendo Switch Combined With Conventional Therapy in People With Acquired Brain Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Isabel Quirosa Galan, Occupational Therapist, MsC, Universidad Rey Juan Carlos
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 291120234382023
Record Dates: First submitted 2024-01-30; First posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Occupational Therapy; Acquired Brain Injury; Adults
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Intervention Model Description: Control Group (CG), which received their usual sessions of conventional therapy sessions, and an Experimental Group (EG), which received therapy with Nintendo Switch plus their conventional therapy sessions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Control Group (CG) which received their usual sessions of conventional therapy.
  Interventions: Procedure: Conventional therapy sessions
- Experimental Group (Experimental): Experimental Group (EG) which received therapy with Nintendo Switch plus their usual sessions of conventional therapy.
  Interventions: Procedure: Conventional therapy sessions plus Nintendo Switch

INTERVENTIONS:
Procedure: Conventional therapy sessions — Conventional sessions are neuropsychology, speech therapy, physiotherapy and occupational therapy treatments. They are based on cognitive stimulation, manipulative dexterity, therapeutic exercise.
  Arms: Control Group
Procedure: Conventional therapy sessions plus Nintendo Switch — Conventional sessions are neuropsychology, speech therapy, physiotherapy and occupational therapy treatments. They are based on cognitive stimulation, manipulative dexterity, therapeutic exercise plus one hour a week of Nintendo Switch.
  Arms: Experimental Group

SUMMARY:
Purpose: to observe the possible benefits produced by conventional therapy through virtual reality with the Nintendo Switch to try to improve motivation and increase the degree of care satisfaction. The aim is to improve postural control in both seated and standing positions and to maintain and improve cognitive capacity.

Material and methods: one group (experimental group) will receive a total of 8 one-hour sessions or 16 half-hour sessions, depending on their individual needs, for 8 weeks using the Nintendo Switch. The other group (control group) will continue to receive their conventional scheduled therapy.

Measures: Abilhand, MEC-Lobo, FIST, Fugl-Meyer, Berg Balance Scale and CSQ-8.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women, over 30 years of age who have suffered an acquired brain injury.
* Mild or moderate cognitive impairment as measured by the MEC-Lobo test (score greater than 23/35).
* Regularly attend some conventional therapy (neuropsychology, physiotherapy or occupational therapy).
* Agree to participate voluntarily by signing the informed consent form.

Exclusion Criteria:

* Present severe cognitive impairment as measured by the MEC-Lobo test (less than 23/35).
* Present aphasia of comprehension or expression.
* Present associated neurodegenerative pathology.
* Present any pathology underlying the acquired brain damage (diabetes, heart disease, COPD, etc.), heart disease, COPD, etc.).
* Voluntarily refuse to participate in the study.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Abilhand | Pre-intervention and post-intervention (up to 1-2 weeks)
  It is an assessment test that measures the degree of difficulty perceived by the patient in performing the 23 activities of daily living.
MEC-Lobo | Pre-intervention and post-intervention (up to 1-2 weeks)
  This is a scale that allows us to evaluate the cognitive status of patients. The lower the score, the greater the cognitive impairment.
Function in Sitting Test (FIST) | Pre-intervention and post-intervention (up to 1-2 weeks)
  It is a scale that assesses the postural control deficits presented by the patient in sedentary position in the event of imbalance, reaching on the floor, etc.
Fugl-Meyer | Pre-intervention and post-intervention (up to 1-2 weeks)
  This scale assesses the patient's motor function, sensory function, muscle balance, range of joint mobility and joint pain.
Berg Balance Scale (BBS) | Pre-intervention and post-intervention (up to 1-2 weeks)
  The scale is used to measure balance mainly in standing position in patients with different types of pathologies.

SECONDARY OUTCOMES:
Client Satisfaction Questionnaire (CSQ-8) | Post-intervention (up to 1-2 weeks)
  Self-administered questionnaire that evaluates the level of satisfaction in relation to the care and quality of care received.

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Quirosa Galan, MsC, Principal Investigator — Universidad Rey Juan Carlos
Locations (1):
- Universidad Rey Juan Carlos, Móstoles, Madrid, Spain